CLINICAL TRIAL: NCT07395908
Title: Comparison of the Effectiveness of Trigeminocervical Complex Peripheral Branch Blockade and Neuromodulation Methods With Peripheral Blood CGRP and PACAP38 Levels in Patients With Chronic Migraine
Brief Title: The Effect of Interventional Procedures on Serum CGRP and PACAP-38 Levels in Chronic Migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Esra Ertilav, Assoc. Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/153
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Migraine Headache; Radiofrequency Ablation; Greater Occipital Nerve Block; Calcitonin Gene-related Peptide; Pacap-38

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients to whom applied radiofrequency (Experimental): For radiofrequency, a 5 cm long RF cannula with a 5 mm active tip is placed in the target under ultrasound guidance, and the needle tip is guided from laterally to medially using an inplane approach to precisely center the nerve. To induce a congruent paresthesia response in the occipital nerve distribution, 50 Hz 1v sensory and 2 Hz 2v motor electrical stimulation was performed with an SMK (Select RF StraightCannula, 100mm, 22G, 10mm active tip SMK-S1010-22) RF electrode. Pulsed radiofrequency (Neurotherm NT1100 / 13001-12) will be applied at 42°C for 240 second
  Interventions: Procedure: Greater occipital nerve Pulse radiofrequency
- patients to whom applied greater occipital nerve block (Active Comparator): The ultrasound probe was placed in a transverse plane 2-3 cm lateral to the Protuberantio Ocipitalis Externa. After visualizing the occipital artery, it was targeted medial to the GON artery. After local anesthesia with 1% lidocaine (skin-subcutaneous), a 21 Gauge 5 cm long needle tip was guided from lateral to medial using an in-plane approach to precisely place it in the center of the nerve for the block (Figure 2). After negative acission, the block was performed with 3 ml of 2% Prilocaine. Supraorbital/supratrochlear nerve block: The ultrasound probe is placed along the supraorbital notch, through the medial third of the supraorbital border. The supraorbital nerve (SON) and the supratrochlear nerve (STN) are located just above its medial border. 2 cc of 2% prilocaine is injected into the target using a 5 cm, 21 gauge needle and inplane technique.
  Interventions: Procedure: Greater occipital nerve block

INTERVENTIONS:
Procedure: Greater occipital nerve Pulse radiofrequency — For radiofrequency, a 5 cm long RF cannula with a 5 mm active tip is placed in the target under ultrasound guidance, and the needle tip is guided from laterally to medially using an inplane approach to precisely center the nerve. To induce a congruent paresthesia response in the occipital nerve distribution, 50 Hz 1v sensory and 2 Hz 2v motor electrical stimulation was performed with an SMK (Select RF StraightCannula, 100mm, 22G, 10mm active tip SMK-S1010-22) RF electrode. Pulsed radiofrequency (Neurotherm NT1100 / 13001-12) will be applied at 42°C for 240 seconds.
  Arms: patients to whom applied radiofrequency
Procedure: Greater occipital nerve block — The ultrasound probe was placed in a transverse plane 2-3 cm lateral to the Protuberantio Ocipitalis Externa. After visualizing the occipital artery, it was targeted medial to the GON artery. After local anesthesia with 1% lidocaine (skin-subcutaneous), a 21 Gauge 5 cm long needle tip was guided from lateral to medial using an in-plane approach to precisely place it in the center of the nerve for the block (Figure 2). After negative acission, the block was performed with 3 ml of 2% Prilocaine. Supraorbital/supratrochlear nerve block: The ultrasound probe is placed along the supraorbital notch, through the medial third of the supraorbital border. The supraorbital nerve (SON) and the supratrochlear nerve (STN) are located just above its medial border. 2 cc of 2% prilocaine is injected into the target using a 5 cm, 21 gauge needle and inplane technique.
  Arms: patients to whom applied greater occipital nerve block

SUMMARY:
The study included 100 patients diagnosed with chronic migraine (CM) who received a diagnosis from the headache clinics of the Neurology Department of Adnan Menderes University Hospitals between May 2025 and May 2026. Inclusion criteria were patients over 18 years of age with chronic migraine. Written informed consent was obtained from all participants; patients with severe systemic diseases, occiput infections or injuries, and allergies to any of the substances used in the injection were excluded. All patients were clinically evaluated (detailed history including personal data, medical history, and migraine treatments used). All patients underwent ultrasound-guided bilateral GON blockade using a portable ultrasound system with a 7-13 MHz multifrequency transducer (ACUSON Juniper Ultrasound System, Siemens, Germany). Blood samples were collected before and one month after the procedure. Samples were collected between 9 and 11 am to avoid the effect of circadian rhythms on CGRP levels. Patients will need to discontinue any anti-inflammatory or analgesic medication within the last 48 hours. A blood sample will be taken from the non-dominant forearm to measure interictal serum CGRP-PACAP38 levels using commercial ELISA kits (Novus Biologicals Inc., USA) according to the manufacturer's instructions. Absorption levels will be measured with a spectrophotometer at a wavelength of 450 nm ± 2 nm. The detection limit for CGRP is 9.3 pg/mL.

DETAILED DESCRIPTION:
Preoperative Visit:

During the preoperative visit, patients' additional illnesses, demographic data, and medication use will be recorded. The patients' NRS (Numerating Rating Scale) score will be recorded. Antebrachial venous blood samples will be taken along with routine samples requested after the outpatient examination.

Intraoperative Nerve Block Procedure:

All procedures were planned to be performed under sterile conditions with ultrasound guidance while the patient was in the prone position.

GON Block: The ultrasound probe was placed in a transverse plane 2-3 cm lateral to the Protuberantio Ocipitalis Externa. After visualizing the occipital artery, it was targeted medial to the GON artery. After local anesthesia with 1% lidocaine (skin-subcutaneous), a 21 Gauge 5 cm long needle tip was guided from lateral to medial using an in-plane approach to precisely place it in the center of the nerve for the block (Figure 2). After negative acission, the block was performed with 3 ml of 2% Prilocaine. Supraorbital/supratrochlear nerve block: The ultrasound probe is placed along the supraorbital notch, through the medial third of the supraorbital border. The supraorbital nerve (SON) and the supratrochlear nerve (STN) are located just above its medial border. 2 cc of 2% prilocaine is injected into the target using a 5 cm, 21 gauge needle and inplane technique.

Intraoperative Pulse Radiofrequency procedure:

For radiofrequency, a 5 cm long RF cannula with a 5 mm active tip is placed in the target under ultrasound guidance, and the needle tip is guided from laterally to medially using an inplane approach to precisely center the nerve. To induce a congruent paresthesia response in the occipital nerve distribution, 50 Hz 1v sensory and 2 Hz 2v motor electrical stimulation was performed with an SMK (Select RF StraightCannula, 100mm, 22G, 10mm active tip SMK-S1010-22) RF electrode. Pulsed radiofrequency (Neurotherm NT1100 / 13001-12) will be applied at 42°C for 240 seconds.

Patients will be observed after the procedure. Patients who do not experience postoperative complications and are mobile will be discharged at 2 hours. Patients may withdraw from the study at any time.

Patients meeting the eligibility criteria will be informed in detail about the procedure. Written and verbal consent will be obtained from the patients.

Post-operative visits:

Venous blood sampling will be performed one month after the procedure, along with routine samples requested after the outpatient examination.

Samples were collected between 9 and 11 a.m. to avoid the influence of circadian rhythms on CGRP levels. Subjects were required to discontinue any anti-inflammatory or analgesic medication in the previous 48 hours. Blood samples were taken from the non-dominant forearm to measure interictal serum CGRP levels using commercial ELISA kits (Novus Biologicals Inc., USA) following the manufacturer's instructions. Absorption levels were measured with a spectrophotometer at a wavelength of 450 nm to 2 nm. The detection limit of the test was considered to be 9.3 pg/ml for CGRP.

For PACAP 38, blood samples were collected into ice-cold glass tubes containing the anticoagulant ethylenediaminetetraacetic acid (EDTA, 12 mg) and the protease inhibitor aprotinin (Trasylol, 1200 IU) and kept at 4°C until centrifuged (2000 rpm for 10 minutes at 4°C). Plasma samples will be stored at -80°C until measured by PACAP-38.

Pain intensity will be assessed using the NRS (Numerical Rating Scale) at 1, 3, and 6 months post-procedure.

The NRS is a pain intensity assessment system based on a system where the individual describes their pain on a scale of 0 (none) to 10 (unbearable pain).

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years of age
2. Having given written consent
3. Patients diagnosed with chronic migraine

Exclusion Criteria:

1. Major psychiatric illness
2. Patients using anticoagulant agents

4. Patients with infection in the procedure area 5. Patients allergic to local anesthetics 6. Pregnant women 7. Patients with cardiac pacemakers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to investigate the effectiveness of nerve block and radiofrequency treatments in patients with chronic migraine using biochemical migraine biomarkers | 1 month
  It was planned to measure venous blood CGRP and PACAP38 levels in patients with chronic migraine before the interventional procedure and one month after the procedure.

SECONDARY OUTCOMES:
The secondary outcome of this study is to compare the effectiveness of nerve block and radiofrequency treatments on chronic pain in patients with chronic migraine. | 6 months
  To evaluate the effectiveness of nerve block and radiofrequency treatments in patients with chronic migraine, a numerical rating scale (NRS) was planned to be applied before the procedure, and at 1, 3, and 6 months after the procedure. An NRS reduction of 50% or more was considered significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Efeler / Aydın, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided